CLINICAL TRIAL: NCT06202417
Title: Fruquintinib in Refractory Metastatic Colorectal Cancer: A Real-world Study
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Director of Colorectal Surgery, Fudan University
Other Study IDs: Fruquintinib real-world
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer; Refractory Colorectal Cancer; Metastatic Colorectal Cancer
Keywords: Fruquintinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; Antineoplastic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- monotherapy group: patients received fruquintinib alone
  Interventions: Drug: Fruquintinib
- combine group: patients administered fruquintinib in combination with chemotherapy or/and anti-PD1 antibodies
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — an oral tyrosine kinase inhibitor (TKI)
  Other Names: PD1 antibodies; chemotherapy drugs

SUMMARY:
Fruquintinib is an oral tyrosine kinase inhibitor (TKI), which improves progression-free survival (PFS) and overall survival (OS) in patients with refractory metastatic colorectal cancer (mCRC). Here, we explore the real-world treatment patterns of fruquintinib in the third- or late-line setting for mCRC in six centers in China.

ELIGIBILITY:
Inclusion Criteria:

(1) histology-confirmed metastatic CRC (mCRC); (2) disease progression on standard therapy with at least two lines of chemotherapy, including fluorouracil, oxaliplatin, and irinotecan with or without biologics such as bevacizumab and cetuximab; (3) fruquintinib administered as salvage treatment; (4) available clinical data.

Exclusion Criteria:

(1) lack of follow-up data; (2) fruquintinib administration as second-line treatment; (3) fruquintinib administration stopped after less than two cycles.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with refractory mCRC and administered fruquintinib from January 1, 2021 to June 31, 2022
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
PFS | Three years
  PFS was calculated from the date of fruquintinib administration to the first observation of disease progression or death
OS | Three years
  OS was defined as the time from fruquintinib administration to death
DCR | During the medication period
  DCR was determined as the proportion of patients who achieved complete response, partial response or stable disease assessed at least 6 weeks after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Contact PI of the study for IPD when publication is online

REFERENCES:
- [Derived] Xu D, Zeng S, Qiu W, Wang G, Qin Z, Liu Y, Zhou S, Zhang Z, Chang W, Feng Q, Xu J. Fruquintinib in refractory metastatic colorectal cancer: a multicenter real-world study. ESMO Open. 2024 Nov;9(11):103702. doi: 10.1016/j.esmoop.2024.103702. Epub 2024 Oct 11. PMID 39395266